CLINICAL TRIAL: NCT05919433
Title: Detection Program for Patients With Primary Biliary Cholangitis Lost in the System
Acronym: RESCAT
Status: Recruiting | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: RESCAT
Record Dates: First submitted 2023-05-29; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with positive AMA and/or ANA anti-gp210/sp100 identified in the hospital database

SUMMARY:
Primary biliary cholangitis (PBC) has been considered a rare disease and its management has been limited by the lack of therapeutic alternatives. PBC is a slowly progressing chronic liver disease characterized by an immune-mediated destruction of the intrahepatic bile ducts, which leads to cholestasis, portal inflammation, and ultimately liver cirrhosis and its associated complications (ascites, portal hypertension, etc), if not treated effectively. Thus, early diagnosis and close management of these patients with PBC is essential. First-line treatment with ursodeoxycholic acid (UDCA) improves liver biochemical parameters, delays histological progression, and increases liver transplant-free survival and overall survival. However, up to 40% of patients are non-responders to UDCA. Obeticholic acid (OCA) is recommended as second-line therapy in combination with UDCA for patients with an inadequate response to UDCA or as monotherapy in cases of UDCA intolerance.

According to current clinical guidelines, the diagnosis of PBC includes a combination of elevated alkaline phosphatase (ALP) levels and the presence of anti-mitochondrial antibodies (AMA) (titer >1:40) and/or anti-nuclear antibodies (ANA) anti-gp210 or anti-sp100. AMA are highly sensitive and specific for PBC and are detected in nearly 95% of PBC patients. A liver biopsy is not necessary unless there is an elevation of ALP without the presence of specific AMA and/or anti-gp210 or anti-sp100 ANA or if coexistence with other liver diseases is suspected (autoimmune hepatitis, hepatic steatosis).

The incidence of PBC has increased in recent years due to an increase in the diagnosis of cases in the initial phases, better awareness in the medical community and the development of more sensitive diagnostic tests. However, up to 31% of patients with PBC are lost without follow-up. The correct identification of patients with PBC is essential so that they can benefit from an adequate treatment and modify disease progression. To date, two studies (one Spanish and one Portuguese) showed that 27% and 45.5% of the patients lost with PBC presented advanced fibrosis, respectively.

The objective of this study is to identify, through computerized data, patients with PBC who may be lost in the system and evaluate their clinical, analytical and demographic characteristics, and in a second phase, provide access to follow-up in specialized consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive AMA and/or with positive ANA anti-gp210 or anti-sp100 identified in the computer databases of each of the participating centers.
* Adults (≥18 years)

Exclusion Criteria:

* Patients with Overlap Syndrome (PBC overlap with Autoimmune Hepatitis (AIH))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified in the database of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients correctly diagnosed with PBC and monitored in specialized health care compared to lost to follow-up PBC patients | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari MútuaTerrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Carey EJ, Ali AH, Lindor KD. Primary biliary cirrhosis. Lancet. 2015 Oct 17;386(10003):1565-75. doi: 10.1016/S0140-6736(15)00154-3. Epub 2015 Sep 11. PMID 26364546
- [Background] Kaplan MM, Gershwin ME. Primary biliary cirrhosis. N Engl J Med. 2005 Sep 22;353(12):1261-73. doi: 10.1056/NEJMra043898. No abstract available. PMID 16177252
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: The diagnosis and management of patients with primary biliary cholangitis. J Hepatol. 2017 Jul;67(1):145-172. doi: 10.1016/j.jhep.2017.03.022. Epub 2017 Apr 18. PMID 28427765
- [Background] Mayo MJ. Mechanisms and molecules: What are the treatment targets for primary biliary cholangitis? Hepatology. 2022 Aug;76(2):518-531. doi: 10.1002/hep.32405. Epub 2022 Mar 10. PMID 35152430
- [Background] Pares A; Leading PBC Group. Practical management of primary biliary cholangitis. Rev Esp Enferm Dig. 2022 Jul;114(7):410-417. doi: 10.17235/reed.2021.8219/2021. PMID 34663072
- [Background] Leung KK, Hirschfield GM. Autoantibodies in Primary Biliary Cholangitis. Clin Liver Dis. 2022 Nov;26(4):613-627. doi: 10.1016/j.cld.2022.06.004. PMID 36270719
- [Background] Olveira-Martin A, Yebra-Carmona J, Amaral-Gonzalez C, Tejedor M, Eiras P, Hernandez-Perez M, Suarez-Cabredo C, Spigarelli-de Rabago I, Suarez-Ferrer C, Morales-Arraez D, Chico I, Diaz-Flores F, Rodriguez R, Llorente S, Molina-Perez E, Hernandez-Guerra de Aguilar MN. Retrieval and treatment of patients with primary biliary cholangitis who are lost in the health system. Rev Esp Enferm Dig. 2021 Nov;113(11):776-779. doi: 10.17235/reed.2021.8174/2021. PMID 34470449
- [Background] Garrido I, Liberal R, Cardoso MJ, Macedo G. The impact of undiagnosed primary biliary cholangitis. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e1027-e1031. doi: 10.1097/MEG.0000000000002268. PMID 34402472